CLINICAL TRIAL: NCT04488679
Title: Clinical and Radiographic Assessment of Platelet Rich Fibrin and Mineral Trioxide Aggregate as Pulp Capping Biomaterials: A Randomized Control Trial
Brief Title: Clinical and Radiographic Assessment of Platelet Rich Fibrin and Mineral Trioxide Aggregate as Pulp Capping Biomaterials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rahma Ahmed Ibrahem Hafiz (Other)
Responsible Party: Sponsor-Investigator, Rahma Ahmed Ibrahem Hafiz, assisstant lecturer- faculty of dentistry- beni suef university, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 111261
Record Dates: First submitted 2020-07-18; First posted 2020-07-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Direct Pulp Capping
Keywords: platelet Rich fibrin , MTA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF along with MTA (Experimental): 5 ml of the participant blood will be drawn into 10 ml test tubes without an anticoagulant and centrifuged immediately .centrifugation will be done using a tabletop centrifuge for 10:12 min at 2700:3000 rounds per minute. The resultant product will exhibit three layers. platelet-poor plasma at the surface, PRF clot in the middle, and red blood cells at the bottom. Sterile tweezers inserted into a test tube to retrieve the PRF clot. The prepared fibrin membrane will be gently packed over the pulp
  Interventions: Other: direct pulp capping
- MTA direct pulp capping (Active Comparator): MTA is primarily calcium oxide in the form of tricalcium silicate, dicalcium silicate and tricalcium aluminate. Bismuth oxide is added for radiopacity, MTA is considered a silicate cement rather than an oxide mixture, a so its biocompatibility is due to its reaction products. MTA elevates the expression of transcription factors, induces dentin bridge formation, possesses biocompatibility9, and sustains a high pH for a longer duration and a close physiochemical seal with dentin that forms an insoluble barrier to prevent microleakag
  Interventions: Other: direct pulp capping

INTERVENTIONS:
Other: direct pulp capping — teeth with exposed pulp during caries removal will be capped either with PRF followed by mta or mta alone directly on exposed pulp, in both groups restoration will be placed over mta
  Other Names: vital pulp therapy

SUMMARY:
eligible carious teeth with exposed pulp by the undergraduate students will be randomly divided into two groups to be treated with direct pulp capping (A), where (A1) represents the comparator group where teeth will be treated with direct application of MTA over the exposed pulp, (A2) represents teeth to be treated with the application of PRF directly over exposed pulp followed by MTA application. clinical and radiographic assessment of tooth vitality, history of pain, pain on percussion, and dentin bridge formation will be performed at baseline, 6 months, and 1 year

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 15:40 years old.
* Patients exhibiting pulp exposure (carious, traumatic, or mechanical) during management of active carious lesions with less than 2 mm of carious exposure.
* Signs and symptoms indicative of pulp vitality, i.e. a positive response to thermal stimulation during a cold test.
* periapical radiograph showing closed apex and normal periapex

Exclusion Criteria:

* Teeth with spontaneous pain or sensitivity to percussion (signs of irreversible pulpitis).
* Teeth with periodontal lesions, internal or external root resorption, calcified canals, mobility of tooth, sinus opening, or abscessed tooth.
* Non restorable tooth.
* Radiographic examination revealed, interrupted or broken lamina dura, widened periodontal ligament space, periapical radiolucency.
* Pulp bleeding that could not be controlled within 10 minutes using 2.5% sodium hypochlorite
* Immune-compromised patients or with systemic medical disorders.
* pregnant females

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 108 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
clinical success rate | 6 months
  pulp vitality by thermal pulp testing
clinical success rate | 6 months
  history of pain
clinical success rate | 6 months
  pain on percussion
clinical success rate | 6 months
  radiographic signs of pulp necrosis and apical periodontitis
clinical success rate | 1 year
  pulp vitality by thermal pulp testing
clinical success rate | 1 year
  history of pain
clinical success rate | 1 year
  no pain on percussion
clinical success rate | 1 year
  radiographic signs of pulp necrosis and apical periodontitis

SECONDARY OUTCOMES:
radiographic assessment of incidence of regenerative dentin (dentin bridge) | 1 year
  assessment of dentin bridge by digital radiography

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Manial, Egypt